CLINICAL TRIAL: NCT01085474
Title: Effect of a Pharmaceutical Intervention on the Level of Control of the Asthmatic Patient
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RES-DUM-2009/1
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
Keywords: Asthma; Pharmaceutical intervention; Effect of a pharmaceutical intervention on the level of control of the asthmatic patient
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 1. Pilot Study: 60 patients (all in the intervention group) 30 patients with intervention A and 30 patients with B intervention)
  Interventions: Other: 1
- 2: Main Study: 600 patients (30 pharmacies control group and 30 pharmacies intervention group, 10 patients per pharmacy)
  Interventions: Other: 2

INTERVENTIONS:
Other: 1 — In the pilot study the objective is to compare 2 different pharmaceutical interventions (A and B) and to assess which one improves disease control, patient adherence and patient knowledge of the medication.
  Groups: 1
Other: 2 — The best intervention used in the pilot study will be chosen and included in the main study.
  Groups: 2

SUMMARY:
Measurement of disease control, treatment adherence and patient knowledge of his/her medication in patients that are receiving a pharmaceutical intervention compared with those patients who receive regular pharmaceutical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given their informed consent and expressed interest in participating in the study
* Asthmatic Patients

Exclusion Criteria:

* Patients with communication difficulties.
* Persons who obtain symbicort but not for their own use.
* Patients with other major diseases: Heart problems, COPD, EMPHYSEMA, lung cancer, AIDS.
* Patients with a respiratory infection.
* Patients with seasonal asthma.
* Pregnant women
* Patients who have previously participated in a health education study in asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 community pharmacies 10 patients per pharmacy
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of the pharmaceutical intervention on the disease control, treatment adherence and patient knowledge of his/her medication using the MEF, treatment adherence and patient knowledge of the medication indicators. | First a Pilot in 3 months and then the final study in 6 months

SECONDARY OUTCOMES:
Compare disease control in patients who know their medication and those who doesn't. | First a Pilot in 3 months and then the final study in 6 months
Compare disease control in patients who comply with their medication with those who doesn't. | First a Pilot in 3 months and then the final study in 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Research Site, Madrid
  - Malaga, Málaga

REFERENCES:
- [Derived] Garcia-Cardenas V, Sabater-Hernandez D, Kenny P, Martinez-Martinez F, Faus MJ, Benrimoj SI. Effect of a pharmacist intervention on asthma control. A cluster randomised trial. Respir Med. 2013 Sep;107(9):1346-55. doi: 10.1016/j.rmed.2013.05.014. Epub 2013 Jun 28. PMID 23810267